CLINICAL TRIAL: NCT00909324
Title: Efficacy, Tolerability and Comfort of 0.3% Hypromellose Eyedrops in the Pre- and Post-Operative Treatment of Patients Undergoing LASIK Surgery
Brief Title: Efficacy, Tolerability, and Comfort of 0.3% Hypromellose Eyedrops in Patients Undergoing LASIK Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CGET980AIN03
Record Dates: First submitted 2009-05-26; First posted 2009-05-28 (Estimated); Results first posted 2011-03-24 (Estimated); Last update posted 2020-08-17 (Actual); Status verified 2020-07

CONDITIONS: Dry Eye
Keywords: Post LASIK dry eye; Pre LASIK dry eye; Hypromellose
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Hypromellose Derivatives

ARMS (2):
- Pre-LASIK 0.3% hypromellose (Experimental)
  Interventions: Drug: Pre-LASIK 0.3% hypromellose
- Post-LASIK 0.3% hypromellose (Active Comparator)
  Interventions: Drug: Post-LASIK 0.3% hypromellose

INTERVENTIONS:
Drug: Pre-LASIK 0.3% hypromellose — Patients self-administered GenTeal eye drops qid (quarter in die, 4 times a day) starting 5 days prior to LASIK surgery and continuing through 1 month after LASIK surgery.
  Arms: Pre-LASIK 0.3% hypromellose
Drug: Post-LASIK 0.3% hypromellose — Patients self-administered GenTeal eye drops qid (quarter in die, 4 times a day) starting on the day of LASIK surgery and continuing through 1 month after surgery.
  Arms: Post-LASIK 0.3% hypromellose

SUMMARY:
This study is designed to assess the tolerability and comfort of peri-operative 0.3% hypromellose eye drops in LASIK surgery patients and to assess whether pre-operative 0.3% hypromellose eye drops add to post-operative comfort in LASIK surgery patients compared to control (no pre-operative lubricant).

ELIGIBILITY:
Inclusion Criteria:

* Age 21 - 35
* Both sexes
* Seeking LASIK surgery at the Refractive Surgery Centre
* Meeting all established criteria for appropriateness for LASIK established by the treating center

Exclusion Criteria:

* Any corneal pathology including scars, prior herpes keratitis, prior corneal transplant
* Any immuno-compromised state including cancer, HIV infection, Hepatitis B or C, or diabetes mellitus
* Requirement for any eye-drops for any reason (eg, dry eye or conjunctivitis) within 3 months from time of enrollment
* Anticipated refusal or inability to undergo planned post-operative visits or assessment
* Failure to meet all established criteria for appropriateness for LASIK

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 170 (Actual)
Dates: Start 2009-08-01 (Actual); Primary Completion 2010-01-01 (Actual); Study Completion 2010-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis India Ltd., Study Director — Novartis India Ltd.
Locations (1):
- Novartis Investigative Site, Delhi, India

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pre-LASIK 0.3% Hypromellose | Post-LASIK 0.3% Hypromellose
Started | 72 | 90
Completed | 72 | 90
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pre-LASIK 0.3% Hypromellose | Post-LASIK 0.3% Hypromellose | Total
Number analyzed (Participants) | 72 | 90 | 162
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26.24 (4.81) | 25.99 (5.06) | 26.10 (4.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 66 | 116
  Male | 22 | 24 | 46

OUTCOME MEASURES:

1. Primary Outcome: Ocular Comfort Level From Baseline to End of Study
Description: Patients rated their ocular comfort on a scale of 0 to 10 on the following parameters: Burning sensation, foreign body sensation, itching, watering of eyes, dryness of eyes, and photophobia. A higher score indicated greater discomfort. A negative change score indicated improvement.
Time Frame: Baseline (Pre-LASIK surgery), Day 1, Day 7 and Day 30 post-LASIK surgery
Population: Intent-to-Treat population: All patients in the study who received study treatment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pre-LASIK 0.3% Hypromellose | Post-LASIK 0.3% Hypromellose
Number analyzed (Participants) | 72 | 90
Units on a scale
  Burning in eyes: Post-LASIK Day 1 | 0.68 (1.18) | 0.84 (1.16)
  Burning in eyes: Day 7 | 0.24 (0.52) | 0.31 (0.54)
  Burning in eyes: Day 30 | 0.08 (0.33) | 0.07 (0.26)
  Foreign body sensation: Post-LASIK Day 1 | 0.94 (1.47) | 1.09 (1.41)
  Foreign body sensation: Day 7 | 0.26 (0.56) | 0.27 (0.55)
  Foreign body sensation: Day 30 | 0.05 (0.29) | 0.09 (0.33)
  Itching: Post-LASIK Day 1 | 0.35 (0.77) | 0.71 (1.21)
  Itching: Day 7 | 0.16 (0.48) | 0.32 (0.68)
  Itching: Day 30 | 0.05 (0.22) | 0.13 (0.42)
  Watering of eyes: Post-LASIK Day 1 | 0.71 (0.94) | 0.71 (0.96)
  Watering of eyes: Day 7 | 0.22 (0.49) | 0.25 (0.49)
  Watering of eyes: Day 30 | 0.10 (0.30) | 0.09 (0.29)
  Dryness of eyes: Post-LASIK Day 1 | 0.82 (1.18) | 1.28 (1.71)
  Dryness of eyes: Day 7 | 0.41 (0.72) | 0.72 (0.98)
  Dryness of eyes: Day 30 | 0.25 (0.60) | 0.49 (0.84)
  Photophobia: Post-LASIK Day 1 | 0.22 (0.54) | 0.41 (0.90)
  Photophobia: Day 7 | 0.09 (0.33) | 0.09 (0.37)
  Photophobia: Day 30 | 0.08 (0.33) | 0.07 (0.26)

2. Secondary Outcome: Tear Breakup Time From Baseline to End of Study
Description: The time required for dry spots to appear on the corneal surface after blinking. Sodium fluorescein dye is added to the eye and the tear film is observed under a slit lamp while the patient avoids blinking until tiny dry spots develop. The longer it takes, the more stable the tear film. A short tear breakup time is a sign of a poor tear film. Generally, >10 seconds is thought to be normal, 5 to 10 seconds marginal, and <5 seconds low (with high likelihood of dry eye symptoms), ie, a shorter time indicates greater eye dryness. A positive change score indicates improvement.
Time Frame: Baseline (Pre-LASIK surgery), Day 1, Day 7 and Day 30 post-LASIK surgery
Population: Intent-to-Treat population: All patients in the study who received study treatment.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Pre-LASIK 0.3% Hypromellose | Post-LASIK 0.3% Hypromellose
Number analyzed (Participants) | 72 | 90
Seconds
  Post-LASIK Day 1 | 14.60 (6.06) | 12.47 (6.20)
  Day 7 | 13.47 (6.22) | 10.84 (3.58)
  Day 30 | 13.63 (5.36) | 12.70 (5.38)

3. Secondary Outcome: Results of Schirmer's Test From Baseline to End of Study
Description: Schirmer's test determines tear production, and whether the eye produces enough tears to keep it moist. A small strip of filter paper is inserted inside the lower eyelid of each eye and the eyes are closed for 5 minutes. The paper is then removed and the length of paper that is moist is measured. A young person normally moistens 15 mm of the paper. The shorter the length of moist paper, the dryer the eyes. A positive change score indicates improvement.
Time Frame: Baseline (Pre-LASIK surgery), Day 1, Day 7 and Day 30 post-LASIK surgery
Population: Intent-to-Treat population: All patients in the study who received study treatment.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Pre-LASIK 0.3% Hypromellose | Post-LASIK 0.3% Hypromellose
Number analyzed (Participants) | 72 | 90
mm
  Left eye: Post-LASIK Day 1 | 19.64 (8.50) | 17.21 (7.10)
  Left eye: Day 7 | 17.68 (9.93) | 17.93 (5.43)
  Left eye: Day 30 | 21.70 (13.01) | 18.77 (7.11)
  Right eye: Post-LASIK Day 1 | 22.65 (7.10) | 13.70 (2.91)
  Right eye: Day 7 | 22.78 (0.49) | 15.25 (0.49)
  Right eye: Day 30 | 22.89 (2.47) | 18.35 (3.83)

ADVERSE EVENTS:
Arm/Group | Pre-LASIK 0.3% Hypromellose | Post-LASIK 0.3% Hypromellose
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/90
Other Adverse Events (participants affected / at risk) | 0/72 | 0/90

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.